CLINICAL TRIAL: NCT03882827
Title: A Prospective, Interventional, Baseline Study In Young Male Subjects Aged From 4 to 9 Years
Brief Title: Natural History of Duchenne Muscular Dystrophy
Status: Recruiting | Type: Observational
Sponsor: Genethon (Other)
Responsible Party: Sponsor
Other Study IDs: GNT-014-MDYF
Record Dates: First submitted 2019-03-18; First posted 2019-03-20 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Duchenne Muscular Dystrophy
MeSH Terms: conditions — Muscular Dystrophy, Duchenne

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood and urine
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Baseline Study on Duchenne Muscular Dystrophy (DMD) in view to collect data on the natural disease course in a cohort in young male subjects aged from 4 to 9 Years over a period of 6 to 36 months using disease appropriate evaluations.

DETAILED DESCRIPTION:
Study duration from FPFV: Q1 2019 to LPLV: Q4 2026

Primary Ojectives:

* To assess the natural disease course using standardized and disease appropriate evaluations in a cohort of young male subjects aged from 4 to 9 years at inclusion and diagnosed for Duchenne Muscular Dystrophy (DMD).
* To record a baseline period prior to rolling over into a gene therapy phase I/II/III clinical study.

Secondary Objectives:

* To identify clinical, imaging and/or laboratory parameters that could be predictive indicators of the disease course in DMD, within the selected range of age.
* To identify the best outcome measure(s) for further clinical trial assessments.

ELIGIBILITY:
Inclusion Criteria:

1. Male
2. 4 to 9 years old inclusive
3. Body-weight ≤ 95th percentile or the BMI scale ≤ 95th percentile (according to validated scale in force in country site).

   Related to the DMD disease:
4. Diagnosis of DMD based upon documented gene testing with detailed genotyping
5. Able to achieve at inclusion and screening visits:

   1. NSAA (North Star Ambulatory Assessment) scale > 18 or ≥ 16 if participant is between 4 and < 5 years old at screening and:
   2. Gowers test < or = 7 sec and/or
   3. 6-Minute Walk Test (6MWT): a distance ≥ 350 meters at inclusion visit (M0)
6. Ongoing corticosteroid therapy or initiation of corticosteroid therapy according to standard of care prior to Screening visit

   Related to the study protocol and ICH/GCP (Good Clinical Practice) requirements:
7. Signed informed consent by at least one parent or both parents or legal guardian representative(s), when applicable and according to the country regulation
8. Affiliated to or a beneficiary of a Health Care scheme (according to country regulation)

   Exclusion Criteria:

   Subject will be excluded from enrolment into the study for any of the following reasons:

   Related to the DMD disease severity:
9. Cardiomyopathy based on physical/cardiological examination and echocardiography with Left Ventricular Simpson biplane Ejection Fraction (LVEF) below 55%
10. Respiratory Assistance: need for either a diurnal and/or a nocturnal ventilation
11. Any co-morbidity (ies) and or previous or planned surgical event(s) which may interfere with DMD natural evolution and or evaluation of outcomes designed to assess DMD Natural History

    Related to specific assessments:
12. Muscle testing: inability to cooperate with
13. MRI: metal implants in regions of interest for the study

    Related to the study protocol and ICH/GCP requirements:
14. Unwilling and/or unable to comply with all the study protocol requirements and/or procedures
15. Previous inclusion to another clinical trial with an Investigational Medicinal Product (IMP), within the 3 months or IMP washout period (whichever is longer) prior to the screening visit of the study
16. Previously treated with a gene therapy drug for DMD, such as:

    * any AAV mediated gene transfer products or any gene editing products in a clinical trial or in a clinical setting,
    * if exons skipping drug was used, the last dose of exon skipping drug within 5 half-lives prior to the screening visit
17. Concomitant participation to any other interventional clinical trial

Ages: 4 Years to 9 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Study Population: * Male
  * 4 to 9 years old inclusive
  * Body-weight ≤ 95th percentile or the BMI scale ≤ 95th percentile (according to validated scale in force in country site).
Sampling Method: Non-Probability Sample
Enrollment: 220 (Estimated)
Dates: Start 2019-12-19 (Actual); Primary Completion 2029-05-30 (Estimated); Study Completion 2029-09-30 (Estimated)

PRIMARY OUTCOMES:
NSAA scale | Screening 36 months
  NSAA scale (age appropriate modified North Star Ambulatory Assessment)
10 Meter Walk/ Run test (10MW/RT) | Screening 36 months
  Time function Test
Raise from floor (RFF) | Screening - 36 months
  Time function test
6 Minutes Walk Test (6 MWT) | Inclusion 36 months
  Motor Function Measurement
Myoset : Myo-grip, -pinch | Inclusion 36 months
  Motor Function Measurement
Stride velocity 95th centile (SV95c) | Inclusion 36 months
  Motor Function Measurement with wearable device (SYDE)
Muscle Imaging Nuclear Magnetic Resonance Imaging (NMRI) | Inclusion 36 months
  Muscle Imaging
Pulmonary Function Test (PFT) | Inclusion 36 months
  Respiratory Function Assessment
ECG - Echocardiography | Inclusion 36 months
  Cardiac Function Assessment
ACTIVLIM | Inclusion 36 months
  Patient Reported Outcome
EQ-5D | Inclusion 36 months
  Questionnaire of Life

CONTACTS AND LOCATIONS:
Overall Officials: Francesco MUNTONI, Pr, Principal Investigator — GOSH LONDON
Locations (15):
- Belgium (3):
  - Centre Hospitalier Universitaire Brugmann, Brussels
  - UZ Leuven, Leuven
  - CHR Hôpital de la Citadelle, Liège
- France (8):
  - University Hospital of Bordeaux, Bordeaux
  - Brest University Hospital Centre, Brest
  - Hopital Femme Mere Enfant, Bron
  - CHU Lille, Lille
  - Hopital la Timone Enfants, Marseille
  - Centre Hospitalier Universitaire - Hôpital Gui de Chauliac, Montpellier
  - Hôpital Armand Trousseau, Paris
  - Hôpital Hautepierre, Strasbourg
- Spain (2):
  - Hospital Sant Joan de Deu Esplugues de Llobregat, Esplugues de Llobregat
  - Hospital La Fe de Valencia, Valencia
- United Kingdom (2):
  - Great Ormond Street Hospital & University College London Hospital, London
  - Institute of Genetic Medicine, Newcastle